CLINICAL TRIAL: NCT06170697
Title: A Single-arm，Single Center，Prospective，Phase II Clinical Study of Camrelizumab Combined With Concurrent Chemoradiotherapy for Short-term Postoperative Progression of Head and Neck Squamous Cell Carcinoma
Brief Title: Advanced First-line Treatment of Short-term Postoperative Progression of Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-OBU-BJ-HNC-II-008
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Immunotherapy; Cisplatin; Drug Therapy; Carboplatin; lobaplatin; nedaplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+（Cisplatin or Carboplatin or Lobaplatin or Nedaplatin）+radiotherapy (Experimental): patients with short-term postoperative progression receive camrelizumab and platin-based chemotherapy concurrent with radiotherapy.
  Interventions: Drug: Camrelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Lobaplatin; Drug: Nedaplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — 200mg, iv, d1, q3w
  Other Names: immunotherapy
Drug: Cisplatin — 80-100mg/m2, iv, q3w, 2-3 cycles in total
  Other Names: chemotherapy
Drug: Carboplatin — AUC 2, iv, q1w, 5-7 cycles in total
  Other Names: chemotherapy
Drug: Lobaplatin — 30mg/m2, iv, q3w, 2-3 cycles in total
  Other Names: chemotherapy
Drug: Nedaplatin — 25-30 mg/m2, iv, q1w, 5-7 cycles in total
  Other Names: chemotherapy
Radiation: Radiotherapy — PGTVp/PGTVnd 66-70Gy/2-2.2Gy/30-35F；PTV1 60Gy/1.8-2.0Gy/30-33F；PTV2 50Gy/1.8-20Gy/25-28F；Start 1-2 weeks after the start of immunotherapy, 1 time before the start of simultaneous chemotherapy, up to 3 times during the concurrent chemoradiotherapy
  Other Names: radiation therapy

SUMMARY:
Every year, about 6% of patients with malignant tumors are diagnosed as head and neck cancer. There are about 650000 new cases and 350000 deaths. A considerable number of patients have simple local recurrence in the short term after operation suggesting that the biological behavior of this kind of tumor is relatively more invasive and the overall prognosis is poor. This project intends to study the efficacy and safety of camrelizumab combined with concurrent chemoradiotherapy for short-term postoperative progression of head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) refers to the general name of squamous cell carcinoma in head and neck organs except nasopharyngeal carcinoma. The main primary sites include oral cavity, oropharynx, hypopharynx, larynx and cervical esophagus. At present, the incidence rate of head and neck squamous cell carcinoma is the sixth most common malignant tumor in the world. Every year, about 6% of patients with malignant tumors are diagnosed as head and neck cancer. There are about 650000 new cases and 350000 deaths, of which squamous cell carcinoma accounts for more than 95%.

In daily clinical work, due to insufficient neck cleaning, slow postoperative incision recovery, long waiting time for treatment, untimely postoperative referral and other reasons, a considerable number of patients have simple local recurrence in the short term after operation (e.g. within 6 months) and before the start of planned adjuvant radiotherapy, so that the purpose of PORT has evolved from initial adjuvant treatment to palliative treatment, It also suggests that the biological behavior of this kind of tumor is relatively more invasive and the overall prognosis is poor. Based on the current clinical and research status, for HNSCC with local regional recurrence in a short time (< 6 months) after operation, both local regional control and remote control must be considered in treatment。 Therefore, this project intends to study the efficacy and safety of camrelizumab combined with concurrent chemoradiotherapy for short-term postoperative progression of head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Sign written informed consent before implementing any test related processes;
* 2.Male or female subjects aged from 18 to 70 years old;
* 3.For head and neck squamous cell carcinoma after standard radical resection and neck lymph node dissection, the number of lymph node dissections is unlimited;
* 4.No neoadjuvant therapy was received before operation and no adjuvant therapy was received after operation;
* 5.Local or regional recurrence has been confirmed by at least 2 radiographs and a pathological diagnosis is not required;
* 6.The time of recurrence was less than 6 months from operation;
* 7.Whole body imaging to rule out distant metastases;
* 8.Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry;
* 9.Adequate haematological, hepatic and renal functions defined by the protocol;
* 10.Estimated life expectancy of more than 1year;
* 11.No history of pD-1 or PD-L1 inhibitor treatment;
* 12.No underlying diseases requiring immunosuppressive therapy;
* 13.PD-L1 status is not required, but PD-L1 IHC detection is recommended;
* 14.Women of reproductive age must undergo a negative urinary pregnancy test within 7 days before starting treatment

Exclusion Criteria:

* 1.The primary site is squamous cell carcinoma of the nasopharynx or skin;
* 2.Previous malignant disease within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, colorectal, breast)；
* 3.Currently participating in intervention clinical research treatment, or receiving other research drugs or using research instruments within 4 weeks before the first administration;
* 4.Previously received anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit T cell receptors;
* 5.Prior organ transplantation, including allogeneic stem-cell transplantation(except corneal transplantation)；
* 6.Known history of allergy to the drug components of this regimen;
* 7.There are multiple factors (e.g. severe renal insufficiency, bone marrow suppression) that influence the chemotherapeutic agent selected by the investigator;
* 8.Before starting treatment, it has not fully recovered from the toxicity and / or complications caused by any intervention;
* 9. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, Active tuberculosis, active hepatitis B (HBV DNA <1000 copy/ml,200 IU/ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method), or co infection of hepatitis B and hepatitis C;
* 10.Accination with live or live/attenuated viruses within 4 weeks of the first dose of camrelizumab and while on trial is prohibited except for administration of inactivated vaccines;
* 11.History of uncontrolled intercurrent illness including hypertension, active infection, diabetes , hereditary bleeding , coagulopathy with a risk of bleedingor, cardiac diseases or symptoms;
* 12.Patients with past and current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-associated pneumonia, and severe impaired lung function may interfere with the detection and management of suspected drug-associated pulmonary toxicity;
* 13.Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy)); The subjects with childhood asthma who had been completely relieved and did not need any intervention or vitiligo in adulthood could be included, but the subjects who needed bronchodilator for medical intervention could not be included;
* 14.Used immunosuppressive drugs within 14 days before the first dose of study drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
1 year Progression-free survival (1y-PFS) | up to 1 years
  Proportion of patients with disease-free survival at 3 years after randomization

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | From the start of randomization to a minimum of 24 months
  Assess ORR, defined as Investigator-assessed CR + PR, per RECIST 1.1.
Disease Control Rate (DCR) | From the start of randomization to a minimum of 24 months
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated
Duration of Response (DoR) | From the start of randomization to a minimum of 48 months
  DoR is defined as the time from the measurement of the first compliance with Cr or pr (whichever occurs first) to the first true recording of disease recurrence or progression.
Overall survival (OS) | From the start of randomization to a minimum of 48 months
  OS is defined as the time (in months) from randomization to the date of death, regardless of the actual cause of the subject's death.
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | From the the first dose of study drug administration up to 28 days after the last dose of study drug administration, assessed up to 2 years
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 28 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, Principal Investigator — Chinese academy of medical science, cancer hospital
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD will be avaliable upon request to PI